CLINICAL TRIAL: NCT06443762
Title: First in Human Study on PET Imaging of Solid Tumors Using an MDM2/MDMX-Specific Probe
Brief Title: First Human Trial of Targeting MDM2/MDMX PET Imaging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023YJZ73
Record Dates: First submitted 2024-05-29; First posted 2024-06-05 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-01

CONDITIONS: MDM2/MDMX Gene Mutation; Nuclear Medicine; Positron Emission Tomography Imaing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group patients who underwent PET scanning with injection probes (Experimental): [68Ga] MDM2/MDMX Peptide PET/CT Imaging: Patients are intravenously injected with prepared and quality-assured [68Ga] MDM2/MDMX Peptide (0.05-0.1 mCi/kg). Imaging is performed 40 minutes to 1 hour post-injection using either the United Imaging uEXPLORER 2m PET/CT or Siemens Biograph m-CT flow PET/CT for whole-body scans, extending from the top of the head to the feet. In cases where conventional imaging reveals indeterminate lesions, delayed imaging is conducted for further differentiation. The patient is positioned supine with calm respiration. The imaging conditions for the head and torso remain as described above. Data are reconstructed using the OSEM method to produce coronal, sagittal, and axial PET and PET/CT fusion images.
  Interventions: Drug: [68Ga] MDM2/MDMX Peptide

INTERVENTIONS:
Drug: [68Ga] MDM2/MDMX Peptide — Utilizing a peptide with high affinity to MDM2/MDMX as the targeting moiety for radiopharmaceuticals, this study explores the diagnostic efficacy of [68Ga] MDM2/MDMX Peptide in patients with malignant tumors exhibiting high MDM2/MDMX expression. This approach not only provides a basis for the early diagnosis of malignant tumors but also facilitates the formulation of effective precision therapy strategies tailored to the tumor's MDM2/MDMX expression profile, particularly for patients with recurrent and metastatic disease.
  [68Ga] MDM2/MDMX Peptide, a novel MDM2/MDMX-targeted molecular probe labeled with 68Ga, utilizes DOTA as a bifunctional chelator for complexing with 68Ga3+. The labeling process is straightforward, allowing for direct use without purification, and demonstrates high in vivo stability.

SUMMARY:
Investigation of the Radiotracer Uptake of [68Ga] MDM2/MDMX Peptide at Lesion Sites in Patients with Malignant Tumors, and Evaluation of the Capability of [68Ga] MDM2/MDMX Peptide to Detect Overexpression of MDM2/MDMX in Tumor Patients, Particularly Those with Recurrent or Advanced Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 75 years, both males and females are eligible;
2. Participants must meet the following criteria for blood routine and liver/kidney function tests: Complete blood count: WBC ≥ 4.0 × 10^9/L or neutrophils ≥ 1.5 × 10^9/L, platelets ≥ 100 × 10^9/L, hemoglobin ≥ 90 g/L; prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal (ULN); liver and kidney function: Total bilirubin ≤ 1.5 times the upper threshold limit (ULT), ALT/AST ≤ 2.5 ULN or ≤ 5 ULT for participants with liver metastasis, alkaline phosphatase (ALP) ≤ 2.5 ULN (if bone or liver metastases are present, ALP ≤ 4.5 ULN); Blood urea nitrogen (BUN) ≤ 1.5 × ULT, serum creatinine (SCr) ≤ 1.5 × ULT;
3. Normal cardiac function;
4. An expected survival of ≥ 12 weeks;
5. Good follow-up compliance;
6. According to RECIST 1.1 criteria, there must be at least one measurable target lesion;
7. Women of childbearing age (15-49 years) must have a negative pregnancy test conducted within 7 days prior to enrollment; patients of childbearing potential must agree to use effective contraceptive methods to ensure they do not conceive during the study and for three months after examinations;
8. Patients recommended for PET/CT evaluation for tumor diagnosis and staging by a clinician;
9. Participants must fully understand the study and voluntarily participate, and must sign an informed consent form.

Exclusion Criteria:

1. Severe abnormalities in liver and kidney function as well as hematological parameters;
2. Patients who are planning a pregnancy;
3. Pregnant or lactating women;
4. Individuals unable to lie flat for thirty minutes;
5. Individuals who refuse to participate in this clinical study;
6. Individuals suffering from claustrophobia or other psychiatric disorders;
7. Other conditions deemed by the researchers as unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
SUV | 1 hour and 2 hours after drug injection
  Standardized Uptake Values (SUV) of [68Ga] MDM2/MDMX Peptide at various time points within the imaging window for target lesions or suspected tumor lesions in subjects with solid tumors or suspected solid tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided